CLINICAL TRIAL: NCT03568201
Title: Application de l'oxymétrie Dynamique et Des Index de Pression Pour le Diagnostic Des Plicatures Iliaques du Sportif
Brief Title: Systolic Ankle arteriaL Pressure and Transcutaneous oximetrY During a TURTLE Test in Athletes
Acronym: SALTY-TURTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018 A01046/ 49
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2020-08

CONDITIONS: Iliac Kinking
Keywords: Diagnosis; Peripheral artery disease; Sports
MeSH Terms: conditions — Disease; Peripheral Arterial Disease | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Intervention Model Description: transcutaneous oximetry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Patients suspected of iliac kinking will have a transcutaneous oximetry test during hip flexion
  Interventions: Diagnostic Test: Transcutaneous oximetry
- controls (Sham Comparator): Healthy asymptomatic athletes will have a transcutaneous oximetry test during hip flexion
  Interventions: Diagnostic Test: Transcutaneous oximetry

INTERVENTIONS:
Diagnostic Test: Transcutaneous oximetry — Measurement of TcpO2 on calves and chests. Calculation of the DROP index (decrease from rest of oxygen pressure)on both calves.

SUMMARY:
Aim of the study is to test the feasibility of transcutaneous oxygen pressure (TcPO2) recording in the diagnosis of iliac kinking in 20 patients with suspected of endofibrosisoriliackinking and 40 asymptomatic control heathy subjects

DETAILED DESCRIPTION:
Patients suspected of PES and healthy controls after detailled explanation of the protocol will have a recording of tcpO2 on both calves and will perform a series of thigh flexion in the standing position.

ELIGIBILITY:
Inclusion Criteria:

- Age over 18 years Insurance company affiliation Symptoms consistent with iliac kinking (patients) or absence of symptoms (controls)

Exclusion Criteria:

* Refuse to participate Exclusion period from another protocole Non affiliation to the French healthcare system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Presence of a significant DROP decrease | 1 hour
  Comparison of DROP value between PES patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, MD, PhD, Principal Investigator — University hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided